CLINICAL TRIAL: NCT04963179
Title: PREvention of Intrauterine Adhesion After Adhesiolysis With Novel Tri-block deGradable Polymer Film.
Acronym: PREG2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Womed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PREG2
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Asherman Syndrome; Intrauterine Adhesion
Keywords: Asherman Syndrome; Intrauterine adhesion; Hysteroscopy; Adhesiolysis; Adhesion prevention; Infertility
MeSH Terms: conditions — Gynatresia; Infertility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Womed Leaf (Experimental): IUA prevention: The novel intrauterine barrier film (Womed Leaf) is inserted immediately after completion of the hysteroscopic adhesiolysis
  Interventions: Device: Womed Leaf
- Control (No Intervention): No IUA prevention - no placebo after adhesiolysis

INTERVENTIONS:
Device: Womed Leaf — Womed Leaf™ device is composed of a uterine anti-adhesion film pre-loaded inside a flexible inserter.
  Womed Leaf™ is inserted in the uterine cavity by the gynecologist surgeon as a film folded into a 5 mm diameter flexible inserter. Once released, the film will unfold and swell into the uterine cavity to keep uterus walls separated. It is degraded and discharged naturally through the cervix and vagina.
  Arms: Womed Leaf

SUMMARY:
PREG2 is a randomized controlled trial that aims to evaluate efficacy in preventing intrauterine adhesion recurrence after hysteroscopic adhesiolysis of a novel intrauterine barrier film named Womed Leaf

DETAILED DESCRIPTION:
PREG2 is a prospective, multi-center, randomized, controlled, two arm clinical study. The objective is to evaluate the efficacy of Womed Leaf in preventing intrauterine adhesion recurrence after adhesiolysis compared to adhesiolysis alone.

The study will be performed on women with moderate or severe adhesions (AFS score >=5) scheduled for adhesiolysis. Indeed, the risk of intrauterine adhesion is very high (up to 60%) in this population of patients.

A follow-up diagnostic hysteroscopy will be performed 6-8 weeks after the adhesiolysis procedure to determine the presence and severity of IUAs according to the American Fertility Society and European Society of Gynecologic Endoscopy classification systems of adhesions. Fertility-related outcome will include live pregnancy at 1 year, 2 years and 3 years and will be reported as secondary endpoints. 154 women are planned to be included in the PREG2 study.

ELIGIBILITY:
Inclusion Criteria:

* Women with moderate or severe intrauterine adhesions according to the AFS classification, i.e AFS score >=5, confirmed by hysteroscopy right before adhesiolysis
* Scheduled for hysteroscopic adhesiolysis
* Age above or equal to 18
* Subjects who are willing to provide a written informed consent.
* Subjects who can comply with the study follow-up (second look hysteroscopy) and other study requirements
* Subjects who agree to refrain from intercourse or use a reliable form of barrier contraception to prevent unintended pregnancy until the follow-up hysteroscopy.
* Subjects who agree to avoid all intrauterine devices (IUDs) until the follow-up hysteroscopy.

Exclusion Criteria:

Pre-operative criteria

* Post menopause
* Pregnant (confirmed by a positive pregnancy test) or lactating
* Abnormal uterine cavity according to ESHRE classification I to V such as unicornis, bicornis, septate, duplex
* Known or suspected endometrial hyperplasia
* History of cervical or endometrial cancer
* Active pelvic infection or history of pelvic peritonitis
* History of endometrial ablation
* Known contraindication or hypersensitivity to Womed Leaf component
* Current participation in another clinical investigation that has not yet received the primary endpoint.
* Any other condition that makes participation in the study contrary to the patient's best interests.

Intra-operative criteria, post adhesiolysis:

* Perforation during adhesiolysis
* Uterine depth < 5cm or > 10cm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (15):
- Gent UZ, Ghent, Belgium
- China (3):
  - Guangdong Maternal and Child Health Hospital, Guangzhou
  - Women's Hospital School Of Medicine Zhejiang University, Hangzhou
  - The Obstetrics & Gynecology Hospital Affiliated to Fudan University, Shanghai
- Gynprenatal, Ostrava, Czechia
- France (5):
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - CHU de Lille, Lille
  - Hopital La Conception, Marseille
  - CHU Lariboisière, Paris
  - Clinique Mutualiste La sagesse, Rennes
- Italy (2):
  - A.O.U Federico II, Napoli
  - Aso Mauriziano Umberto I, Torino
- Spain (2):
  - Hospital Clinic Barcelonna, Barcelona
  - Ramon y Cajal Hospital, Madrid
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the result that will be reported in an article and study protocol may be made available to researchers who provide a methodologically sound proposal, immediately after article publication and during 5 years
Supporting Information: Study Protocol
Time Frame: immediately after article publication and during 5 years
Access Criteria: researchers who provide a methodologically sound proposal

REFERENCES:
- [Derived] Fernandez H, Miquel L, Sroussi J, Weyers S, Munmany M, Luo X, Kovar P, Wang Y, Zizolfi B, Surbone A, Delporte V, Moratalla E, Sauvan M, Perrini G, Sui L, Mara M. Effectiveness of degradable polymer film in the management of severe or moderate intrauterine adhesions (PREG-2): a randomized, double-blind, multicenter, stratified, superiority trial. Fertil Steril. 2024 Dec;122(6):1124-1133. doi: 10.1016/j.fertnstert.2024.07.020. Epub 2024 Jul 22. PMID 39048019

RESULTS

PARTICIPANT FLOW:
Groups:
- Womed Leaf: IUA prevention: The novel intrauterine barrier film (Womed Leaf) is inserted immediately after completion of the hysteroscopic adhesiolysis
  Womed Leaf: Womed Leaf™ device is composed of a uterine anti-adhesion film pre-loaded inside a flexible inserter.
  Womed Leaf™ is inserted in the uterine cavity by the gynecologist surgeon as a film folded into a 5 mm diameter flexible inserter. Once released, the film will unfold and swell into the uterine cavity to keep uterus walls separated during approximately 5 days. It is degraded and discharged naturally through the cervix and vagina in less than 30 days.
Period: Overall Study
Arm/Group | Womed Leaf | Control
Started | 75 | 85
Completed | 71 | 82
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Control: No IUA barrier - No placebo
- Total: Total of all reporting groups
Arm/Group | Womed Leaf | Control | Total
Number analyzed (Participants) | 75 | 85 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (5.2) | 35.9 (5.1) | 35.5 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 85 | 160
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 71 | 80 | 151
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 15 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 18 | 33
  White | 47 | 52 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 5 | 6 | 11
  Czechia | 13 | 13 | 26
  China | 11 | 13 | 24
  Italy | 4 | 1 | 5
  France | 37 | 42 | 79
  Switzerland | 1 | 2 | 3
  Spain | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Efficacy - IUA Severity
Description: Change of AFS score between pre-adhesiolysis and second-look hysteroscopy (AFS) score
  The scale used to assess the severity of intrauterine adhesions is the American Fertility Society score. It is a 12 points composite score that adds-up 3 subcomponents: - Extend of adhesions (1 = less than 1/3 of the uterine cavity involved with adhesions to 4 = more than 2/3 of the uterine cavity involved with adhesions),
  * Type of adhesions (1 = Filmy adhesions to 4 = dense adhesions)
  * Menstrual pattern (0= normal to 4 = amenorrhea).
  The final score allows the following prognostic classification:
  1-4 = mild disease, 5-8 = moderate disease 9-12 = severe disease
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Population: The modified ITT (mITT) included all randomized patients, apart from 3, who were incorrectly randomized prior to, rather than after, their baseline hysteroscopy and were then excluded for not fulfilling the preset operative criteria without contributing any effectiveness data to the study.
  There were 163 patients randomized in total. The mITT population includes 163-3= 160 patients; 75 in the Womed Leaf group and 85 in the Control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Womed Leaf: Womed Leaf resorbable barrier is inserted right after adhesiolysis.
- Control: No IUA barrier
Arm/Group | Womed Leaf | Control
Number analyzed (Participants) | 75 | 85
score on a scale | 5.2 (2.8) | 4.2 (3.2)

2. Primary Outcome: Safety - Adverse Events
Description: Adverse events up to second look hysteroscopy.
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Womed Leaf | Control
Number analyzed (Participants) | 77 | 86
Participants | 6 | 3

3. Secondary Outcome: High-responder Rate
Description: Percentage of patients who have improved from severe to mild adhesions or from severe to no adhesions or from moderate to no adhesions
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change of "Extent of Cavity Involved" Component
Description: Average of AFS score component "extent of cavity involved"
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change in "Extent of Cavity Involved" Component Between Post-adhesiolysis and Second Look Hysteroscopy
Description: Average of AFS score component "extent of cavity involved"
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

6. Secondary Outcome: AFS Score
Description: Average of AFS score
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Change of Extent of IUA AFS Score Component
Description: Average of the change of the AFS score component "Extent of IUA"
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Change of Type of IUA AFS Score Component
Description: Average of the change of the AFS score component "type of IUA"
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Menstrual Pattern AFS Score Component
Description: Average of the change of the AFS score component "Menstrual Pattern"
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Percentage of Patients Who Have Mild Adhesions or no Adhesion
Description: Percentage of patients who have AFS < 5
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Freedom From IUA
Description: Rate of patients who don't have adhesion
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

12. Secondary Outcome: ESGE Stage
Description: Rate of ECGE stage
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Level of Post-operative Pain
Description: Level of post-operative pain on a numeric rating scale, with 0 = no pain and 10 = the worst pain.
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Level of Discomfort Related to Vaginal Discharge
Description: Level of discomfort related to vaginal discharge on a numeric rating scale, with 0 = no discomfort and 10 = extremely disturbing
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Timing of Vaginal Discharge
Description: Timing of vaginal discharge as recalled by the patient
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

16. Secondary Outcome: Duration of the Vaginal Discharge
Description: Duration of the vaginal discharge as recalled by the patient
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

17. Secondary Outcome: Qualitative Description of the Vaginal Discharge
Description: Qualitative description of the vaginal discharge as recalled by the patient
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

18. Secondary Outcome: Change of Menstrual Pattern
Description: Change of menstrual pattern
Time Frame: At second look hysteroscopy between 4 and 8 weeks, 1 year, 2 years
Reporting Status: Not Posted

19. Secondary Outcome: Reintervention Rate
Description: Reintervention rate, during second look hysteroscopy or scheduled later up to one year
Time Frame: At second look hysteroscopy or scheduled later up to one year
Reporting Status: Not Posted

20. Secondary Outcome: Number of Adhesiolysis Procedures
Description: Number of adhesiolysis procedures after second look to one year
Time Frame: After second look to one year
Reporting Status: Not Posted

21. Secondary Outcome: Pregnancy Rate
Description: Pregnancy rate defined as presence of foetal sac or heartbeat by ultrasound at 1 year and 2 years, whether spontaneous or IVF
Time Frame: 1 year, 2 years, 3 years
Reporting Status: Not Posted, anticipated posting 2027-03

22. Secondary Outcome: Live Birth Rate
Description: Live birth rate at 1 year and 2 years
Time Frame: 1 year 2 years, 3 years
Reporting Status: Not Posted, anticipated posting 2027-03

23. Secondary Outcome: Pregnancy Complication Rate
Description: Pregnancy complication rate
Time Frame: 3 years
Reporting Status: Not Posted, anticipated posting 2027-03

24. Secondary Outcome: Time to Pregnancy
Description: Time to pregnancy (i.e. time between the second look hysteroscopy and pregnancy start)
Time Frame: 3 years
Reporting Status: Not Posted, anticipated posting 2027-03

25. Secondary Outcome: IUA Severity According to Chinese Scoring System
Description: IUA severity according to Chinese scoring system (for patients enrolled in China only)
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

26. Secondary Outcome: Responder Rate
Description: Percentage of patients with an improvement of one clinical category i.e from Severe to Moderate or from Moderate to Mild
Time Frame: At second look hysteroscopy between 4 and 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Womed Leaf | Control
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/86
Other Adverse Events (participants affected / at risk) | 6/77 | 3/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Womed Leaf (N=77) | Control (N=86)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Uterine perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervix disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT04963179/Prot_SAP_000.pdf